CLINICAL TRIAL: NCT06787274
Title: Improving Health Equity by Understanding Preferences in Telehealth Abortion
Brief Title: Research on Equity in Abortion Care by TeleHealth
Acronym: REACH
Status: Recruiting | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: Ibis Reproductive Health (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: 23-39122; R01HD110659 (NIH)
Record Dates: First submitted 2024-04-05; First posted 2025-01-22 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Abortion in First Trimester; Abortion Early; Abortion; Attempted
Keywords: health equity; medication abortion; telehealth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- In-person via established clinic: People seeking or who have received in-person medication abortion care through an established clinic.
- Telehealth via established clinic: People seeking or who have received telehealth medication abortion care through an established clinic. A telehealth medication abortion involves a remote clinical consultation to confirm medical eligibility with medications delivered by mail
- Telehealth through other online services or searches: People seeking or who have received telehealth medication abortion care through an online service
- In-person through online search: People seeking or who have received in-person abortion services through online searches

SUMMARY:
This study will examine the ways in which telehealth for reproductive healthcare affects timing, costs, and follow-up care; whether telehealth reaches people in areas with greater health inequities; and the attributes of telehealth that patients want. Study surveys will be administered to interested, eligible participants: 2,000 patients seeking abortion care will complete the study, comprising of 2 groups: patients seeking medication abortion care either (1) in-person or (2) via telehealth. This project will address how telehealth services can be optimized for people of color, low-income people, and immigrants to increase digital inclusion and health equity.

DETAILED DESCRIPTION:
Given the novelty of telehealth abortion services and new abortion bans, there is a critical need for research on the role of telehealth for abortion to expand equitable abortion access among groups historically marginalized in healthcare. Outside of abortion care, telehealth appears to 1) bridge geographic disparities,2) facilitate language translation,3) provide privacy and safety for immigrants with varying legal statuses, 4) decrease patient costs, and 5) require less time off work or school. At the same time, telehealth services could exacerbate inequities if patients lack technology, internet connectivity, or digital literacy. Because abortion is overregulated and highly stigmatized, research on telehealth for abortion is vital. The investigators hypothesize that telehealth is associated with several benefits compared to in-person abortion care, but is not yet reaching people in areas with greater health inequities who need these innovations most. This research can also inform the policies in states that are considering ways to support people in banned states.

ELIGIBILITY:
Inclusion Criteria:

* Must be currently or about to be obtaining medication abortion care through in-person or telehealth services

Exclusion Criteria:

* Not currently or about to be obtaining medication abortion care through in-person or telehealth services

Ages: 14 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Participants who have recently received or are currently seeking medication abortion, either through in-person or telehealth services will be able to participate on this study. Up to 1,000 participants will be enrolled through established clinics that offer in-person and telehealth services (500 in-person clinic patients; 500 telehealth patients). Up to 1,000 participants will be enrolled online via Google Ads or other online outreach methods (500 in-person clinic patients and 500 telehealth patients).
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2025-02-12 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Determine the ways in which telehealth services affect timing and time to care by comparing in-person and telehealth patients | Baseline
  Descriptive statistics for the elapsed days from the first pregnancy test to 1) date of the decision to have an abortion, 2) date of first contact with the clinic, 3) date of medication receipt, and 4) date mifepristone (the first medication) was ingested.
Determine the ways in which telehealth services affect costs by comparing in-person and telehealth patients | Baseline and 1 week
  Report of 1) out-of-pocket costs for the abortion and 2) the costs of related expenses, including transportation, childcare, lost work, and other expenses.
Determine the ways in which telehealth services affect follow-up care by comparing in-person and telehealth patients | 1 week
  The incidence of unplanned in-person follow-up visits to a clinician, emergency room, or other facility, between participants in the telehealth and in-person groups using logistic regression models.

SECONDARY OUTCOMES:
Investigate the patient preferences for different aspects of telehealth for abortion care among historically marginalized groups | Baseline and 1 week
  We will conduct a discrete choice analysis to understand participant preferred choices for hypothetical delivery alternatives to telehealth abortion.
Investigate the barriers in telehealth for abortion care in historically marginalized groups | Baseline and 1 week
  The barriers to hypothetical delivery alternatives to telehealth abortion between participants in the telehealth and in-person groups using a discrete choice model

CONTACTS AND LOCATIONS:
Overall Officials: Ushma Upadhyay, PhD, MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- Advancing New Standards in Reproductive Health (ANSIRH), Oakland, California, United States

IPD SHARING:
Plan to Share IPD: No